CLINICAL TRIAL: NCT03130140
Title: Macroscopic On-site Quality Evaluation of Biopsy Specimens to Improve the Diagnostic Accuracy During EUS-guided FNA Using a 19-gauge Needle for Solid Lesions: a Multicenter Prospective Randomized Controlled Study
Brief Title: MOSE to Improve the Diagnostic Accuracy During EUS-guided FNA Using a 19-gauge Needle for Solid Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Charing Chong, MD, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2015.511
Record Dates: First submitted 2017-04-19; First posted 2017-04-26 (Actual); Last update posted 2018-12-06 (Actual); Status verified 2018-12

CONDITIONS: Solid Tumor

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Macroscopic on-site evaluation (Active Comparator): EUS-FNA perform with a 19-gauge needle with macroscopic on-site evaluation.
  Interventions: Procedure: Macroscopic on-site evaluation
- Control (Sham Comparator): EUS-FNA perform with a 19-gauge needle with conventional techniques.
  Interventions: Other: Control

INTERVENTIONS:
Procedure: Macroscopic on-site evaluation — Macroscopic on-site evaluation: any aspirated material on a glass slide for inspection of the presence of a macroscopic visible core (MVC). Length of MVC will be measured to determine the adequacy of that puncture.
  Arms: Macroscopic on-site evaluation
Other: Control — Conventional EUS-FNA
  Arms: Control

SUMMARY:
The technique of macroscopic on-site evaluation (MOSE) has recently been advocated for estimating the adequacy of a core specimen for histological diagnosis during EUS-FNA using a 19-gauge needle. How it compares to the conventional technique of tissue acquisition during EUS-FNA is uncertain.

The objective of this study is to evaluate the quantity and quality of tissue, and the diagnostic ability of MOSE when compared with the conventional combined histologic-cytologic analysis.

DETAILED DESCRIPTION:
To evaluate the quantity and quality of tissue, and the diagnostic ability of MOSE when compared with the conventional combined histologic-cytologic analysis in a randomized controlled study.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients (aged between 18 and 80 years) referred for EUS-guided tissue acquisition for intestinal or extra-intestinal solid lesions more than 2cm in the largest diameter would be included.

Exclusion Criteria:

* Patients with coagulopathy, altered anatomy, contraindications for conscious sedation, pregnancy and those who cannot provide informed consent would be excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Estimated)
Dates: Start 2016-02-26 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic yield: Proportion of patients with adequate tissue for diagnosis obtained by EUS FNA | 4 weeks
  proportion of patients with adequate tissue for diagnosis obtained by EUS FNA

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chong CCN, Lakhtakia S, Nguyen N, Hara K, Chan WK, Puri R, Almadi MA, Ang TL, Kwek A, Yasuda I, Doi S, Kida M, Wang HP, Cheng TY, Jiang Q, Yang A, Chan AWH, Chan S, Tang R, Iwashita T, Teoh AYB. Endoscopic ultrasound-guided tissue acquisition with or without macroscopic on-site evaluation: randomized controlled trial. Endoscopy. 2020 Oct;52(10):856-863. doi: 10.1055/a-1172-6027. Epub 2020 Jun 4. PMID 32498098